CLINICAL TRIAL: NCT06132529
Title: Biomarker Signature to Predict the Persistence of Post-traumatic Headache
Brief Title: A Study to Evaluate Biomarker Signature to Predict the Persistence of Post-traumatic Headache
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Arizona State University (Other)
Responsible Party: Principal Investigator, Catherine (Cat) Chong, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005203; R61NS113315 (NIH)
Record Dates: First submitted 2023-10-25; First posted 2023-11-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Post-Traumatic Headache; Healthy
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Magnetic Resonance Imaging; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Post-Traumatic Headache Group: Subjects diagnosed with having post-traumatic headache complete an MRI, speech sample, and electronic daily headache diary.
  Interventions: Diagnostic Test: Brain Magnetic Resonance Imaging (MRI) Scan; Other: Speech Sample; Other: Electronic Daily Headache Diary
- Healthy Control Group: Subjects identified as health and not having any headaches will complete an MRI and speech sample.
  Interventions: Diagnostic Test: Brain Magnetic Resonance Imaging (MRI) Scan; Other: Speech Sample

INTERVENTIONS:
Diagnostic Test: Brain Magnetic Resonance Imaging (MRI) Scan — Imaging of the brain
Other: Speech Sample — Recorded reading aloud of pre-written words and sentences
Other: Electronic Daily Headache Diary — Headache diary to provide information about headaches experience that day.
  Groups: Post-Traumatic Headache Group

SUMMARY:
The purpose of this research study is to develop a model to help distinguish patients at high-risk for developing persistent post-traumatic headache from patients who experience headache recovery. Researchers will do this by comparing the brain images, clinical data, and speech of healthy controls to people who have been diagnosed with post-traumatic headache.

ELIGIBILITY:
Inclusion Criteria:

* Post-traumatic headache (PTH) and persistent post-traumatic headache (PPTH) will be diagnosed using the ICHD-3 diagnostic criteria for PTH attributed to mild traumatic brain injury (concussion).
* For patients with PTH, only patients with new onset of PTH without history of PPTH will be included in the study.
* A personal history of prior concussion and history of migraine are allowed according to ICHD-III diagnostic criteria.
* Tension-type headaches on three or fewer days per month is allowed for healthy control subjects.

Exclusion Criteria:

* History of moderate or severe traumatic brain injurie (TBI).
* Prior history of gross anatomical change on imaging.
* Contraindication to MRI, including but not limited to severe claustrophobia and/or presence of ferrous materials in the body.
* Women who are pregnant, or believe that they might be pregnant. Although there are no known contraindications or risks associated with pregnancy and MRI, we will exclude pregnant women or women who believe that there might be a chance that they are pregnant.
* History of concussion or more severe TBI.
* History of migraine or other headaches.
* The diagnosis for PTH and PPTH will be verified by Dr. Schwedt (co-investigator) a board-certified physician in Neurology and Headache Medicine. Presence of concussion will be verified using the Ohio State University TBI Identification Method, a standardized questionnaire assessing the lifetime history of TBI for an individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected through a multi-site collaboration between the Mayo Clinic Headache and Concussion Clinics in Arizona and the Phoenix VA Health Care System.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Prediction of post-traumatic headache recovery | 6 years
  Using questionnaires and fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chong, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - VA Health Care System, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20502645